CLINICAL TRIAL: NCT06907615
Title: An Open-label, Multi-center, Global Phase II Clinical Study to Evaluate the Efficacy and Safety of HLX43 (Anti-PD-L1 ADC) in Subjects With Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Phase II Clinical Study to Evaluate HLX43 in Subjects With Advanced Non-small Cell Lung Cancer (NSCLC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Collaborators: Henlius USA Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLX43-NSCLC201
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-04

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- HLX43 DOSE 1 (2.0 mg/kg) (Experimental): Patients with good tolerability and well controlled disease will receive the treatment once every 3 weeks (Q3W), Until disease progression, initiation of a new anti-tumor therapy, death, emergence of intolerable toxicity, or withdrawal of informed consent (whichever occurs first)
  Interventions: Drug: HLX43 DOSE 1 (2.0 mg/kg)
- HLX43 DOSE 2 (2.5 mg/kg) (Experimental): Patients with good tolerability and well controlled disease will receive the treatment once every 3 weeks (Q3W), Until disease progression, initiation of a new anti-tumor therapy, death, emergence of intolerable toxicity, or withdrawal of informed consent (whichever occurs first)
  Interventions: Drug: HLX43 DOSE 2 (2.5 mg/kg)

INTERVENTIONS:
Drug: HLX43 DOSE 1 (2.0 mg/kg) — Dose 1; 2.0 mg/kg; HLX43 is an anti-PD-L1 monoclonal antibody conjugated with a novel high potency DNA topoisomerase I (topo I) inhibitor, with a drug-antibody-ratio (DAR) of 8.
  Arms: HLX43 DOSE 1 (2.0 mg/kg)
Drug: HLX43 DOSE 2 (2.5 mg/kg) — Dose 2; 2.5 mg/kg; HLX43 is an anti-PD-L1 monoclonal antibody conjugated with a novel high potency DNA topoisomerase I (topo I) inhibitor, with a drug-antibody-ratio (DAR) of 8.
  Arms: HLX43 DOSE 2 (2.5 mg/kg)

SUMMARY:
The study is being conducted to to explore the reasonable dosage and evaluate the efficacy, safety and tolerability of HLX43 (Anti-PD-L1 ADC) in Patients with Advanced Non-small Cell Lung Cancer (NSCLC)

DETAILED DESCRIPTION:
This study is an open-label phase II clinical study to explore the reasonable dosage and evaluate the efficacy, safety and tolerability of HLX43 (Anti-PD-L1 ADC) in Patients with advanced non-small cell lung cancer (NSCLC). In this study, eligible subjects will be randomized at 1:1 ratio, and the patients will be administered with HLX43 at different doses via intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

* Have a full understanding of the study content, process, and possible adverse reactions before the study, and sign the informed consent form (ICF); voluntarily participate in the study; be able to complete the study as per protocol requirements;
* Aged ≥ 18 years at the time of signing the ICF, male or female;
* Histologically or cytologically confirmed, locally advanced (stage IIIB/IIIC) or metastatic (stage IV) NSCLC not suitable for radical treatment (complete surgical resection, concurrent/sequential radio-chemotherapy) according to the Union for International Cancer Control and the American Joint Committee on Cancer (AJCC) TNM staging system (8th edition), and should meet the following criteria:

  1. Subjects without actionable genomic alterations (AGAs):

     * Subjects with non-squamous NSCLC must have documented negative test results for EGFR and ALK alterations. If no prior test results for EGFR and ALK are available, subjects must undergo EGFR and ALK testing at the study site. For subjects with squamous NSCLC, EGFR and/or ALK testing is not required prior to enrollment if their status is unknown;
     * No other known actionable genomic alterations, such as ROS1, NTRK, BRAF, MET exon 14 skipping, and RET;
     * Prior standard treatment failure of ≥ 1 line, including at least anti-PD-(L)1 antibody and platinum-based chemotherapy;
  2. Subjects with AGAs:

     * Previous test results confirming the presence of one or more actionable genomic alterations;
     * Prior standard treatment failure of ≥ 1 line, including at least targeted therapy for driver gene alterations (patients with EGFR mutations must be previously treated with EGFR inhibitors) and platinum-based chemotherapy;
* At least one measurable lesion as per RECIST 1.1 within 4 weeks prior to randomization;
* Subjects who agree to provide archived tumor tissue specimens that meets the testing requirements (either from the most recent surgery or biopsy, preferably within 2 years) or agree to undergo a biopsy to collect tumor tissue for PD-L1 expression testing;
* The following conditions must be met in terms of the time of the first administration of the investigational product: at least 3 weeks (or 5 half-lives of the drug, whichever is shorter) from the previous major surgery, medical device treatment, locoregional radiotherapy (except for palliative radiotherapy for bone lesions), cytotoxic chemotherapy, immunotherapy, or biological product therapy; at least 2 weeks from the previous hormone therapy or small molecular targeted therapy; at least 1 week from the administration of the traditional Chinese medicine for anti-cancer indications or minor surgery; and recovery of treatment-induced AEs to Grade ≤ 1 (CTCAE v5.0, except for Grade 2 peripheral neurotoxicity and alopecia);
* ECOG PS score of 0-1 within 1 week prior to randomization;
* Life expectancy > 3 months;
* Adequate organ functions as confirmed by laboratory tests within 1 week prior to randomization (no blood transfusions or treatment with granulocyte colony-stimulating factor is allowed within 14 days prior to the first dose)
* Male and female subjects with child-bearing potential must agree to use at least one highly effective contraception method during the study and within at least 6 months after the last dose of the investigational product; female subjects of childbearing age must be negative for pregnancy test within 7 days prior to enrollment.

Exclusion Criteria:

* Histologically or cytologically confirmed tumor containing components of small cell lung cancer, neuroendocrine carcinoma, or sarcomatoid carcinoma;
* Prior treatment with any medication targeting topoisomerase I, including chemotherapy or ADCs;
* Radical radiation therapy within 3 months prior to the first dose;
* History of any second malignancy within 2 years prior to randomization, except for early-stage malignancies (carcinoma in situ or stage I tumors) that have received radical treatment, such as non-melanoma skin cancer, cervical carcinoma in situ, localized prostate cancer, ductal carcinoma in situ of the breast, and papillary thyroid carcinoma;
* History of adverse events leading to permanent discontinuation of immunotherapy, or occurrence of ≥ Grade 2 immune-related pneumonitis or myocarditis during prior immunotherapy;
* Presence of uncontrollable pleural effusion, pericardial effusion, or ascites requiring repeated drainage;
* Presence of spinal cord compression or clinically active metastases to central nervous system (referring to untreated or symptomatic metastases, or metastases requiring corticosteroids or anticonvulsants to control associated symptoms), carcinomatous meningitis. Subjects who have previously received treatment for brain metastases (such as whole brain radiotherapy or stereotactic brain radiotherapy) may be eligible, provided that they are clinically stable for at least 4 weeks with no imaging evidence of brain metastasis progression;
* Subjects with current or prior history of clinically significant pulmonary impairment due to pulmonary comorbidities, including but not limited to any underlying lung disease (e.g., pulmonary embolism within 3 months prior to the first dose, severe asthma, severe chronic obstructive pulmonary disease, restrictive lung disease, interstitial pneumonia, pneumoconiosis, drug-related pneumonitis, and pleural effusion within 3 months prior to the first dose), any autoimmune, connective tissue, or inflammatory disease that may involve the lungs (i.e., rheumatoid arthritis, Sjogren's syndrome, sarcoidosis), prior pneumonectomy that may interfere with the detection and management of suspected drug-related pulmonary toxicity, or history of with radiation pneumonitis within 6 months;
* Patients with any poorly-controlled cardiovascular and cerebrovascular clinical symptoms or diseases, including but not limited to: (1) NYHA Class II or greater heart failure or left ventricular ejection fraction (LVEF) < 50%; (2) unstable angina pectoris; (3) myocardial infarction or cerebrovascular accident within 6 months (except lacunar infarction, slight cerebral ischemia, or transient ischemic attack); (4) poorly controlled arrhythmia (including QTc intervals ≥ 470 ms) (QTc intervals are calculated by Fridericia's formula); (5) poorly-controlled hypertension (systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg after active treatment);
* Patients with active systemic infectious diseases requiring intravenous antibiotics within 2 weeks prior to randomization;
* Patients who have used moderate or potent CYP2D6 or CYP3A inhibitors or inducers within 2 weeks prior to randomization;
* Patients who have received systemic corticosteroids (prednisone > 10 mg/d or equivalent dose of similar drug) or other immunosuppressants within 2 weeks prior to randomization; Except: patients treated with topical, ocular, intra-articular, intranasal, and inhaled corticosteroids; short-term prophylactic use of corticosteroids for contrast agents, etc.;
* Patients with known active or suspected autoimmune diseases. Patients with autoimmune-related hypothyroidism and receiving thyroid hormone replacement therapy and those with type 1 diabetes mellitus controlled with insulin therapy are eligible to be enrolled;
* Patients who have received live vaccine or live attenuated vaccine within 4 weeks prior to randomization;
* Patients who are known to have anaphylaxis to macromolecular protein preparations/monoclonal antibodies or are allergic to any component in the formulation of the investigational product;
* Patients with active tuberculosis;
* Patients with a history of immunodeficiency, including human immunodeficiency virus (HIV)-positive or other acquired or congenital immunodeficiencies, or history of organ transplantation;
* Patients with active HBV or HCV infection or HBV/HCV co-infection;
* Pregnant or lactating women;
* Patients who are not suitable for participating in this clinical study due to any clinical or laboratory abnormalities or other reasons as assessed by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2028-04-20 (Estimated); Study Completion 2028-06-04 (Estimated)

PRIMARY OUTCOMES:
ORR | From date of the first dose of study drug until the date of death from any cause, assessed up to 24 months
  Objective response rate (ORR) (assessed by the Independent Radiology Review Committee [IRRC] as per RECIST v1.1).

SECONDARY OUTCOMES:
ORR | From date of the first dose of study drug until the date of death from any cause, assessed up to 24 months
  Objective response rate (ORR) (assessed by the investigator as per RECIST v1.1).
PFS | From date of the first dose of study drug until the date of death from any cause, assessed up to 24 months
  Progression-free survival (PFS) (assessed by the IRRC and the investigator as per RECIST v1.1)
OS | From date of the first dose of study drug until the date of death from any cause, assessed up to 24 months
  Overall survival (OS)
Incidence and severity of adverse events (AEs) | From date of the first dose of study drug until the date of death from any cause, assessed up to 24 months
  severity determined according to National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] Version [v] 5.0, vital signs and clinical laboratory test results

CONTACTS AND LOCATIONS:
Overall Officials: Jie He, Dr, Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Jie Wang, Dr, Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Fred Hirsch, Dr, Study Chair — Mount Sinai Health System
Locations (2):
- MD Anderson Cancer Hospital, Houston, Texas, United States
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China